CLINICAL TRIAL: NCT02985450
Title: A Prospective Study of Hepatitis B Virus (HBV) Immunity and Hepatitis B Vaccination in Patients With Non Alcoholic Fatty Liver Disease (NAFLD) in Canada
Brief Title: A Prospective Study of HBV Immunity and HBV Vaccination in Patients With NAFLD in Canada
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: REB16-0274
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2018-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Hepatitis B; Vaccine Reaction
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis B | interventions — Engerix-B; twinrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs will be cryopreserved to assess HBV specific T and B cell responses.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Engerix-B — Hepatitis B Vaccine
  Other Names: Twinrix

SUMMARY:
(1) Due to missed childhood vaccination programs, the majority of adult patients with NAFLD in Canada do not have immunity to hepatitis B. (2) Adults with NAFLD who receive the HBV vaccine have reduced immunogenic responses in the setting of obesity (i.e., protective anti-HBs titres). Aims: (1) To determine the sero-prevalence of immunity against hepatitis B in a cohort of prospectively evaluated adult NAFLD patients. (2) To prospectively determine HBV vaccine responses (anti-HBs titres) in adult NAFLD patients.

DETAILED DESCRIPTION:
The hepatitis B virus (HBV) is truly a global human pathogen that affects at least 2 billion people worldwide including ~240 million chronic hepatitis B (CHB) carriers that are at risk for end-stage liver disease. The diagnosis of CHB is confirmed by the persistence of the HBV surface antigen (HBsAg) in serum for >6 months. However, a latent form of HBV infection known as occult hepatitis B infection (OBI) characterized by low-level viremia (i.e., HBV DNA < 200 IU/ml) despite undetectable serum HBsAg has been described with unclear clinical consequences.

A safe and effective HBV vaccine has been available for ~3 decades and consists of recombinant HBsAg which contains the major viral antigenic epitopes and induces a protective neutralizing antibody to HBsAg (anti-HBs) response in >85% of children vaccinated. Canada is a low HBV-endemic region and in Alberta, and Ontario, public health uses maternal screening for HBsAg to identify babies at-risk for CHB. Thus, all infants born to HBsAg (+) mothers are given passive-active immunoprophylaxis with hepatitis B immune globulin (HBIG) and the HBV vaccine within 12 hours of birth, as well as 2 doses at ~2 and ~6 months of age. Testing of the infants for anti-HBs is recommended at 9 months to ensure immunity. In the late 1990's, a universal HBV childhood vaccination program was initiated in all Canadian provinces and jurisdictions. In Alberta and in Ontario, school-age children are scheduled to receive the 3-dose HBV vaccine series in grade 5. However there remain a significant proportion of adult Canadians (i.e., born before 1985) who missed childhood vaccination programs. Although current guidelines recommend that certain high-risk populations receive hepatitis B immunization, appropriate identification and compliance is generally much lower in adults compared to children.

According to the most recent Canadian Association for the Study of Liver Disease guidelines, all adults with diabetes, as well as all patients with chronic liver disease should receive the hepatitis B vaccine. The basis for these recommendations are two-fold, (1) diabetics may be at risk of blood-borne virus (BBV) exposure through contact with contaminated blood glucose monitoring devices and (2) diabetic patients are at increased risk of the metabolic syndrome and the development of non-alcoholic fatty liver disease (NAFLD). The improvement in blood glucose monitoring devices, and increased knowledge has reduced the risk of HBV exposure in patients with diabetes. Further, the investigators' initial seroepidemiological survey of acute HBV outbreaks in Alberta revealed a decreasing prevalence in diabetic patients. Therefore the main incentive for HBV vaccination in diabetics is due to the concomitant risk of the metabolic syndrome and advanced liver disease due to NAFLD. There is limited data on HBV vaccination in NAFLD patients. Further studies are required in a North American adult (Canadian population).

The investigators propose that adults with NAFLD should undergo comprehensive screening for hepatitis B immunogenicity, in addition to screening for infection, and catch up or booster vaccinations should be administered to non-immunized patients with confirmatory immunity testing thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-60 years of age, who provide signed informed consent
* Diagnosis of NAFLD/NASH according to expert assessment (by imaging, TE, abnormal lab tests and/or liver biopsy)
* No evidence of prior infection or immunity to hepatitis B (negative HBsAg, anti-HBs, anti-HBc).

Exclusion Criteria:

* Subjects < 18 years of age,
* Subjects who refused vaccination
* Have documented immunity / prior exposure to hepatitis B (i.e., positive for ant-HBs, anti-HBc, HBsAg)
* Pregnancy
* HIV-positive
* Decompensated cirrhosis (i.e., Child-Pugh Class B or C) due to impact on immune response.
* Subjects >60 y will be excluded, due to effect of age and reduced response to HBV vaccination.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: NAFLD patients will be recruited from large tertiary liver clinics in Canada
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-08; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Coffin, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with non-alcoholic fatty liver disease (NAFLD), without prior exposure to hepatitis B or hepatitis B vaccine. Recruitment period was August 2016-March 2020.
Pre-assignment Details: No significant events were noted. 7 patients were lost to follow-up.
Groups:
- HBV Vaccine Cohort: Of 82 participants, all received the HBV vaccine. Vaccines were not blinded as patients were followed as standard of care. We followed the product monograph for TWINRIX and Engerix vaccines.
Period: Overall Study
Arm/Group | HBV Vaccine Cohort
Started | 82
Completed | 75
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: 7 patients lost to follow-up.
Groups:
- HBV Vaccine Cohort: Of 82 participants, all received the HBV vaccine. Vaccines were not blinded as patients were followed as standard of care.
Arm/Group | HBV Vaccine Cohort
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (8.7)
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 82
BMI (body mass index) [Mean (Standard Deviation); unit: kg/m^2] | 33.6 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Anti-HBs Titres (IU/L)
Description: to determine how NAFLD-associated metabolic risk factors and liver inflammation / fibrosis affects vaccine response
Time Frame: 1 month after completion of the vaccine series
Population: Anti-HBs levels were compared between two groups: low and high-risk obesity patients with NAFLD.
Measure: Mean (Standard Deviation); unit: Anti-HBS IU/L
Groups:
- BMI < 35: 40 patients with BMI < 35
- BMI > 35: 28 patients with BMI > 35
Arm/Group | BMI < 35 | BMI > 35
Number analyzed (Participants) | 40 | 28
Anti-HBS IU/L | 642 (68.2) | 385 (79)
Statistical Analysis 1: Comparison: BMI < 35 vs BMI > 35; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 513.5, Standard Deviation 73.6 — Anti-HBs levels difference: high risk obesity group - low risk obesity group NAFLD patients

2. Primary Outcome: Assessment of Memory T Cells and HBsAg-specific-proliferation of CD3 + CD4+ TH Cells
Description: to determine how NAFLD-associated metabolic risk factors and liver inflammation / fibrosis affects vaccine response. Fresh (or cryopreserved in 4 patients) PBMC (~106) were labeled with 1 μM carboxyfluorescein-diacetate-succinimidyl-ester. Labeled PBMC were stimulated with 5 μg HBsAg) in RPMI 1640 with 10% FBS and 2mmol/L glutamine. Anti-CD3 (1 μg/mL) and anti-CD28 (5 μg/mL) stimulated cells served as a positive control.
  Unstimulated DMSO-treated cells were used as negative controls. Cells were cultured in triplicates and plates incubated at 37 °C with 5% CO2 for ~8 days. Cell proliferation was assessed on day 8. SI was calculated as % CFSE low cells in stimulated cells / % CFSE low cells in the unstimulated control46. SI> 3 was considered positive for HBsAg-specific proliferation. Cells were stained using the memory T-cell panel and analyzed by flow-cytometry
Time Frame: 1 month after completion of the vaccine series
Population: 17 patients with BMI < 35 and 14 patients with BMI > 35 for PBMC analysis.
Measure: Mean (Standard Deviation); unit: Stimulation index
Groups:
- BMI < 35: 17 patients with BMI < 35 and PBMCs collected for analysis.
- BMI > 35: 14 patients with BMI > 35 and PBMCs collected for analysis.
Arm/Group | BMI < 35 | BMI > 35
Number analyzed (Participants) | 17 | 14
Stimulation index | 5.1 (0.68) | 3.1 (0.62)

ADVERSE EVENTS:
Time Frame: Each patient was assessed with 18 months of their baseline visit. Antibodies titers were assessed within 3 months after their last hepatitis vaccine dose.
Arm/Group | HBV Vaccine Cohort
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT02985450/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT02985450/ICF_001.pdf